CLINICAL TRIAL: NCT02771678
Title: Estimating the Loss in Quality of Life Associated With an Asthma Related Crisis Event (ESQUARE)
Brief Title: Estimating Quality of Life in People With Asthma
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/EE/0023
Record Dates: First submitted 2016-05-05; First posted 2016-05-13 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2016-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma: All participants will have an asthma-related crisis event due to an asthma exacerbation that resulted in A&E attendance and/or hospital admission.

SUMMARY:
The aim of this project is to estimate the quality of life for people with asthma and specifically the loss in quality of life associated with an asthma-related crisis event (accident and emergency (A&E) attendance or admission).

DETAILED DESCRIPTION:
Asthma is a serious respiratory condition which causes shortness of breath, chest tightness and wheezing. Quality of life can have an impact on asthmatics due to such symptoms. Previous studies capture quality of life at specific time points (e.g. baseline, 1 month, 3 months), and the assumption of a steady improvement is made. However, these assumptions and time points could miss an asthma event in between. Therefore, the investigators aim to provide a more accurate estimation of the loss in quality of life by following participants over an 8 week period from when the participants have attended A&E or been admitted to hospital following an asthma attack. This will be done by using different quality of life methods, and analysed by calculating the difference between the quality of life scores from A&E attendance / hospital admission and follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years old and over
* Has asthma alone, or asthma with Chronic Obstructive Pulmonary Disease (COPD) or asthma with a respiratory infection
* Speaks English
* Not in need of help from carer / guardian to complete questionnaires
* Not hypoxemic
* Not participated in the study before
* Able to give informed consent

Exclusion Criteria:

* Younger than 18 years old
* Does not speak English
* Has participated in the study before
* Remains hypoxemic despite oxygen therapy
* Impaired capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients who have an asthma-related crisis event (attended A&E or have been admitted to hospital).
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
EuroQol 5 Dimensions 5 Level (EQ-5D-5L) | Once a week from baseline until week 8
  A generic quality of life questionnaire
Asthma Quality of Life Questionnaire (AQLQ) | Once a month from baseline to week 8
  A disease-specific quality of life questionnaire
Peak flow and asthma symptom diary | Every day from baseline to week 8
  Assessment of peak expiratory flow and asthma symptoms
Time Trade-Off | Once a month from baseline to week 8
  Assessment of quality of life. Completed at Norfolk and Norwich University Hospital only.

SECONDARY OUTCOMES:
Productivity Questionnaire | Week 4
  Assessment of time lost from work, study or activities from having an asthma exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Christina-Jane Crossman-Barnes, BSc, MSc, Principal Investigator — University of East Anglia; Andrew Wilson, MD FRCP, Principal Investigator — University of East Anglia
Locations (3):
- United Kingdom (3):
  - Norfolk and Norwich University Hospital, Norwich, Select A County
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen Elizabeth Hospital Birmingham, Birmingham

REFERENCES:
- [Derived] Crossman-Barnes CJ, Sach T, Wilson A, Barton G. Estimating loss in quality of life associated with asthma-related crisis events (ESQUARE): a cohort, observational study. Health Qual Life Outcomes. 2019 Apr 11;17(1):58. doi: 10.1186/s12955-019-1138-5. PMID 30971261